CLINICAL TRIAL: NCT01881542
Title: Comparison of the Standard 24-hour Urine Protein With Shorter Collection Periods for the Diagnosis of Preeclampsia
Brief Title: Standard 24-hour Urine Protein vs Shorter Period for Diagnosis of Pre-eclampsia
Acronym: PET and urine
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Raed Salim, MD, HaEmek Medical Center, Israel
Other Study IDs: 0157-12-EMC
Record Dates: First submitted 2013-06-11; First posted 2013-06-19 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2022-08

CONDITIONS: Preeclampsia
Keywords: preeclampsia; proteinuria; urine collection
MeSH Terms: conditions — Pre-Eclampsia; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background and project rationale:

Preeclampsia is a common complication of pregnancy, affecting 6-8% of all pregnancies and constitutes a leading cause of maternal morbidity and mortality. Preeclampsia is liable to endanger the lives of both the gravida and the fetus, particularly if treatment is initiated inappropriately or in an untimely fashion.

Diagnosis of preeclampsia is dependent on the finding of proteinuria, determined as being over 300mg of protein in a 24 hours urine sample. However, urine collection spanning 24 hours sometimes constitutes a "bottleneck", extending the time to diagnosis of preeclampsia. Additionally, the collection of urine for 24 hours entails a degree of discomfort, requiring that the woman be in proximity to for collection vessel, and increases the length of her hospital admission.

The use of an abbreviated test may permit diagnosis and treatment in a more timely fashion. Similarly, the ability to exclude the diagnosis more rapidly could reduce length of hospital stay and consumption of the health system's limited resources. Further, a shorter test may reduce the discomfort associated with the 24-hour test and thus increase compliance.

Previous research has suggested that briefer tests correlate with the traditional 24 hour urine collection, however these studies were based on small study populations.

Research Objective:

To validate a brief and rapid test for the diagnosis of urinary protein excretion.

To assess whether, in women with suspected preeclampsia, a difference exists between protein excretion during the daytime and at night.

Methods:

Urine collection will be performed on pregnant women admitted for investigation of suspected preeclampsia, with volumes recorded and samples taken at 6, 12 and 24 hour intervals for assessment of urinary protein content. As such, a comparison will be made between the protein excretion after 6 and 12 hours with that over a full 24 hour period; in addition, comparison will be made between daytime and nighttime urinary protein excretion. The results will allow for assessment of whether a shorter test can substitute the full 24 hour collection in the diagnosis of preeclampsia; results of women who are shown to not suffer from preeclampsia will be used to assess whether a short test can rule out the disease. Additionally a urine sample for protein/creatinine ratio will be examined and correlated with results of the different collection periods.

DETAILED DESCRIPTION:
Literature review and project rationale:

Preeclampsia is a common complication of pregnancy, affecting 6-8% of all pregnancies and constitutes a leading cause of maternal morbidity and mortality. Preeclampsia is liable to endanger the lives of both the gravida and the fetus, particularly if treatment is initiated inappropriately or in an untimely fashion.

The diagnosis of preeclampsia is based on findings of raised blood pressure (over 140/90mmHg) and the presence of proteinuria. The accepted means of measuring proteinuria is by 24-hour urine collection, with a pathological value defined as 300mg or greater in the 24 hour period. When the proteinuria is greater than 5000mg in 24 hours, the pr-eclampsia is classified as severe and is further endangers the lives of the expectant mother and fetus and often results in early delivery.

Diagnosis and assessment of severity of preeclampsia require a timely situation assessment. Urine collection spanning 24 hours sometimes constitutes a "bottleneck", extending the time to diagnosis of preeclampsia. Additionally, the collection of urine for 24 hours entails a degree of discomfort, requiring that the woman be in proximity to for collection vessel, and increases the length of her hospital admission.

The use of an abbreviated test may permit diagnosis and treatment in a more timely fashion. Similarly, the ability to exclude the diagnosis more rapidly could reduce length of hospital stay and consumption of the health system's limited resources. Further, a shorter test may reduce the discomfort associated with the 24-hour test and thus increase compliance.

Previous research has shown that 8-hour urine collection does indeed produce results paralleling the 24-hour collection, and recent research also demonstrates concordance between 12-hour and 24-hour urine collections. That said, both these studies were based on small sample populations, fewer than 100 women. Another study of women with preeclampsia showed good correlation between the results of urinary protein in samples collected over 12 hours at night and those collected over 12 hours during daytime.

Research Assumptions:

1. urine collection for a period of time less than 24 hours will reflect the degree of urinary protein excretion.
2. urine collection for a period of time less than 24 hours will constitute an alternative test for 24-hour urine collection, the accepted diagnostic test today.

Research Objective:

To validate a brief and rapid test for the diagnosis of urinary protein excretion.

To assess whether, in women with suspected preeclampsia, a difference exists between protein excretion during the daytime and at night.

Methods:

Urine collection is to be performed on every pregnant admitted for investigation of suspected preeclampsia. After 6, 12 and 24 hours samples of the collected urine will be taken for protein concentration assessment. Quantitative urinary protein will be established according to urinary protein concentration and collected urine volume. Results of the tests after 6 and 12 hours will be compared to the final results after 24 hours, that being the test of choice for diagnosis of proteinuria in preeclampsia and thus the test that will determine management (according to department protocol).

Women for whom preeclampsia has been ruled out (viz, those who underwent investigation following raised BP but without a finding of proteinuria) will serve to assess the ability of a short urine collection to rule out proteinuria and, as such, preeclampsia.

So as to assess whether there is a difference between results of daytime urinary protein excretion and those at night, the urine collection will be performed in two vessels as follows:

1. 8:00am - beginning of urine collection
2. 2:00pm, vessel 1 - recording of collected urine volume, removal of a 10mL sample of urine for protein concentration testing.
3. 8:00pm, vessel 1 - recording of total collected urine volume, removal of a 10mL sample of urine for protein concentration testing.

   at this point urine collection will be continued in the second vessel
4. 8:00am the following morning, vessel 2 - recording of collected urine volume as of 8:00pm (the previous 12 hours), removal of a 10mL sample of urine for protein concentration testing.
5. contents of the two vessels are mixed, 24 hour urine volume recorded and a 10mL sample taken, this being the sample that will establish the result of the 24 hour urine collection.

Additionally a urine sample for protein/creatinine ratio will be examined and correlated with results of the different collection periods.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* age 18-55 years
* blood pressure >140mmHg systolic or >90mmHg diastolic

Exclusion Criteria:

* known renal disease
* urinary tract infection
* spontaneous labor or need to induce labor within the first 24 hours of admission

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women admitted for assessment of suspected preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2023-07 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
to validate a shorter urine collection time for assessment of proteinuria | one year
  urine collection over 6 and 12 hours to compare with results of the official 24 hours urine collection for proteinuria in the investigation of suspected preeclampsia
To examine if a shorter urine collection time for assessment of proteinuria is comparable to the standard 24 hours | one year

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, M.D., Principal Investigator — haemek medical center
Locations (1):
- HaEmek Medical Center, Afula, Israel

REFERENCES:
- [Background] Tun C, Quinones JN, Kurt A, Smulian JC, Rochon M. Comparison of 12-hour urine protein and protein:creatinine ratio with 24-hour urine protein for the diagnosis of preeclampsia. Am J Obstet Gynecol. 2012 Sep;207(3):233.e1-8. doi: 10.1016/j.ajog.2012.06.010. Epub 2012 Jun 11. PMID 22939731
- [Background] Shennan AH, Redman C, Cooper C, Milne F. Are most maternal deaths from pre-eclampsia avoidable? Lancet. 2012 May 5;379(9827):1686-7. doi: 10.1016/S0140-6736(11)60785-X. Epub 2011 Dec 14. No abstract available. PMID 22177535
- [Background] Adelberg AM, Miller J, Doerzbacher M, Lambers DS. Correlation of quantitative protein measurements in 8-, 12-, and 24-hour urine samples for the diagnosis of preeclampsia. Am J Obstet Gynecol. 2001 Oct;185(4):804-7. doi: 10.1067/mob.2001.117302. PMID 11641655
- [Background] Kieler H, Zettergren T, Svensson H, Dickman PW, Larsson A. Assessing urinary albumin excretion in pre-eclamptic women: which sample to use? BJOG. 2003 Jan;110(1):12-7. PMID 12504929